CLINICAL TRIAL: NCT04229238
Title: Nutrition and Medication Management in Home-dwelling Older Adults. Study I: Nutritional Status and Medication Treatment in Home-dwelling Older Adults. A Cross-sectional Study
Brief Title: Nutritional Status and Medication Treatment in Home-dwelling Older Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Collaborators: The Norwegian Research Fund for General Practice (Unknown)
Responsible Party: Principal Investigator, Mari Fiske, Principal Investigator, University of Oslo
Other Study IDs: 2017/12883-1
Record Dates: First submitted 2019-12-27; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Malnutrition; Aged; Polypharmacy
Keywords: Nutritional status; Polypharmacy; Home-dwelling; Potentially inappropriate medication use
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home-dwelling older adults: Older adults (70 +) receiving regular health care from the home nursing service. Setting is two rural municipalities in southern Norway.

SUMMARY:
The project "Nutrition and Medication management in home-dwelling older adults" consist of two separate studies witch are described in the same study protocol. This is the first study in this Project. The second study is described separately; Identification: 2017/12883-2

Malnutrition is common in older adults. The causes are many and include adverse drug effects. Loss of appetite, nausea, or dry mouth are adverse drug effects, which may contribute to malnutrition. Knowledge about possible relations between drug treatment and nutritional status is scarce.

The objectives of the project is to describe nutritional status, drug treatment and the prevalence of potentially inappropriate medication in home-dwelling elderly receiving home care service in two Norwegian municipalities.

DETAILED DESCRIPTION:
Recruitment by a the home nurse service. An informed content from the participant (or a close relative for those not able to give an informed consent) is required. A nurse will visit the participants and ask for information about six items concerning: food intake, weight loss, mobility, psychological stress, neuropsychological problems. The height and weight will be measured. A photo of the medicine prescription card will be taken. The investigators have created an online solution for collection of these sensitive data, including photos of the medication prescription card.

The data will automatically be stored in a secure database at the University of Oslo (TSD), for further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Home-dwelling
* Be admitted to home-nursing service, every second week or more often.
* Age 70 or older
* Medication administrated by home nursing service.
* Informed consent by patient or close relative (next of kin)

Exclusion Criteria:

• Patient or next of kin denies inclusion

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults (70 +) receiving regular health care from the home nurse service. Setting is two rural municipalities in southern Norway.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | week 1
  By use of Mini Nutritional Assessment Short Form (MNA-SF).Maximum value 14, minimum value 0. 0 -7 points indicates malnutrition. 8-11 points indicate risk for malnutrition. 12-14 points indicates well nourished. The higher score a better outcome.
Potential Inappropriate medication | week 1
  Prevalence of potential Inappropriate medication due the Norwegian General Practise Nursing home( NORGEP) criteria.
  A: Single criteria; Regular use should be avoided. B: Combination criteria; Combinations to avoid C: Deprescribing (discontinue) criteria: Need for continued use should be reassessed: See Protocol page 19-20; Attachment 1.
Drugs with high risk for causing nausea, loss of appetite and dry mouth | week 1
  Prevalence of drugs with high risk for causing nausea, loss of appetite and dry mouth, according to a list we have made( Nause-Appetite-Dry mouth list) see Protocol page 21-23,attachment 2

CONTACTS AND LOCATIONS:
Overall Officials: Jørund Straand, professor, Study Chair — Institute of Health and Society, University of Oslo, Norway
Locations (1):
- University of Oslo, Institute for Health and Society, Department of General Practice, Oslo, Norway

DOCUMENTS (3):
  • Informed Consent Form: Participants (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT04229238/ICF_000.pdf
  • Informed Consent Form: to next of kin (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT04229238/ICF_001.pdf
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT04229238/Prot_002.pdf